CLINICAL TRIAL: NCT02080481
Title: Effect of InfinitiPlusTM Needle Guidance in Ultrasound Guided Regional Anesthesia
Brief Title: Needle Guidance in Ultrasound Guided Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1299
Record Dates: First submitted 2014-02-21; First posted 2014-03-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Elective Knee Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infiniti Plus needle guidance system (Experimental): ultrasound guidance with the InfinitiPlus (TM) needle guidance system
  Interventions: Device: Infiniti Plus needle guidance system
- conventional block needle (Other): ultrasound guidance with a conventional block needle
  Interventions: Device: Conventional block needle

INTERVENTIONS:
Device: Infiniti Plus needle guidance system — The Infiniti Plus needle guidance system is designed to help physicians perform ultrasound guided nerve blocks.
  Arms: Infiniti Plus needle guidance system
Device: Conventional block needle — conventional block needle used for insertion of femoral nerve catheters.
  Arms: conventional block needle

SUMMARY:
An FDA-approved product, InfinitiPlus (TM), is a needle guidance system that has been recently developed to guide clinicians in performing ultrasound guided nerve blocks. This system helps the clinician to align the needle with ultrasound beam while performing an ultrasound guided nerve block. InfinitiPlus (TM) has a unique open channel design allowing efficient needle movement while having improved needle shaft and tip visualization. This is a disposable system specifically designed for improving success rate of ultrasound guided block and patient safety.

This study will be done with patients having elective knee surgery and a femoral nerve block with a catheter. The nerve block procedure will be performed under ultrasound guidance to help improve safety and efficacy of the injection. InfinitiPlus (TM) has been recently developed to try to improve needle guidance in the ultrasound guided nerve block procedure. This study will determine whether femoral nerve block procedures performed under ultrasound guidance with InfinitiPlus (TM) take less time than procedures performed with ultrasound guidance and a conventional block needle. The study will also determine whether the InfinitiPlus (TM) needle reduces the number of times the clinician attempts the procedure, reduces the cost of the procedure, increases the procedure success rate, and improves ultrasound visibility of the needle.

Participants will be randomly assigned to either ultrasound guidance with the InfinitiPlus (TM) needle guidance system or ultrasound guidance with a conventional block needle. After surgery, pain will be rated every 30 minutes for the first 2 hours, then every 4 hours while awake for 24 hours. 24 hours after surgery, participants will be given a survey about pain treatment satisfaction and a questionnaire about recovery.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-85 years old
* Scheduled for elective knee surgery and expected to receive a femoral nerve block and catheter
* Written informed consent

Exclusion Criteria:

* Contraindications to femoral block such as coagulopathy, infection at the needle insertion site and allergy to local anesthetics
* Pregnancy
* Preexisting neuropathy involving the surgical limb

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Turan A, Babazade R, Elsharkawy H, Esa WA, Maheshwari K, Farag E, Zimmerman NM, Soliman LM, Sessler DI. Novel needle guide reduces time to perform ultrasound-guided femoral nerve catheter placement: A randomised controlled trial. Eur J Anaesthesiol. 2017 Mar;34(3):135-140. doi: 10.1097/EJA.0000000000000584. PMID 28009637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Started | 68 | 67
Completed (The patients completed the study were included in the analysis) | 67 | 67
Not Completed | 1 | 0
Not completed — Never received a block. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.6) | 63.8 (9.1) | 64.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 30 | 23 | 53
Intraoperative management strategy [Count of Participants; unit: Participants]
  General anesthesia | 42 | 36 | 78
  Spinal anesthesia | 23 | 31 | 54
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Performing Ultrasound Guided Femoral Nerve Blocks With InfinitiPlusTM Needle Guidance System
Time Frame: time elapsed from beginning the block procedure (after prepping and draping) until the catheter was successfully inserted or the end of the day of surgery.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Number analyzed (Participants) | 67 | 67
seconds | 118 [100 to 150] | 177 [130 to 236]
Statistical Analysis 1: Comparison: Infiniti Plus Needle Guidance System vs Conventional Block Needle; Test type: Superiority or Other; p < 0.001, Regression, Linear; intraoperative management strategy was imbalanced between randomized groups and was adjusted for in the linear regression model; ratio of geometric means = 0.68, 95% CI 2-sided [0.61 to 0.76]

2. Secondary Outcome: Block Failure
Description: Number of patients who had block failure
Time Frame: start of surgery until femoral nerve block completion
Measure: Count of Participants; unit: Participants
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Number analyzed (Participants) | 67 | 67
Participants | 5 | 3
Statistical Analysis 1: Comparison: Infiniti Plus Needle Guidance System vs Conventional Block Needle; Test type: Superiority or Other; p = 0.56, Regression, Logistic; intraoperative management strategy was imbalanced between randomized groups and was adjusted for in the logistic regression model; Odds Ratio (OR) = 1.55, 98.3% CI 2-sided [0.25 to 9.6] — Odds ratio for Infiniti Plus versus conventional needle patients

3. Secondary Outcome: > 1 Block Attempt
Description: Number of block attempts was collected for each patient as > 1 block attempt versus 1 attempt. A block attempt was defined as pulling the block needle back to skin and redirecting it.
Time Frame: from start of block procedure until block placement
Measure: Count of Participants; unit: Participants
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Number analyzed (Participants) | 67 | 67
Participants | 1 | 7
Statistical Analysis 1: Comparison: Infiniti Plus Needle Guidance System vs Conventional Block Needle; Test type: Superiority or Other; p = 0.06, Regression, Logistic — Intraoperative management strategy was imbalanced between groups and adjusted for in the logistic regression model; Odds Ratio (OR) = 0.13, 98.3% CI 2-sided [0.01 to 1.78]

4. Secondary Outcome: Percentage of Time With Perfect Needle Visibility
Description: Percentage of time that perfect needle visibility was visualized on ultrasound.
Time Frame: From start of block procedure until block placement
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Number analyzed (Participants) | 67 | 67
percentage of time | 59 (28) | 55 (24)
Statistical Analysis 1: Comparison: Infiniti Plus Needle Guidance System vs Conventional Block Needle; Test type: Superiority or Other; p = 0.74, Regression, Linear; Intraoperative management strategy was imbalanced between randomized groups and adjusted for in the linear regression model; Mean Difference (Final Values) = 4.4, 98.3% CI 2-sided [-7.7 to 14.6]

ADVERSE EVENTS:
Arm/Group | Infiniti Plus Needle Guidance System | Conventional Block Needle
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes